CLINICAL TRIAL: NCT07146854
Title: EndoForce Post Approval Study
Status: Recruiting | Type: Observational
Sponsor: Phraxis, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 009-034
Record Dates: First submitted 2025-08-21; First posted 2025-08-28 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: End Stage Renal Disease (ESRD)
Keywords: Hemodialysis; Arteriovenous graft
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No

GROUPS / COHORTS (1):
- EndoForce: AV Graft implanted using the EndoForce Connector for Endovascular Venous Anastomosis

SUMMARY:
The goal of this observational study is to collect long-term safety and performance data for the use of the EndoForce System for connecting a hemodialysis graft to a vein in patients with End Stage Renal Disease. This is not an experimental procedure or an experimental therapy. This means that the study device has been approved by the FDA.

ELIGIBILITY:
Inclusion Criteria:

* Patient is ≥18 years of age.
* Patient requires the creation of a vascular access graft for hemodialysis, secondary to a diagnosis of ESRD.
* Patient is able to have the vascular access ePTFE graft placed in an upper arm.
* Patient or his/her legal guardian understands the study and is willing and able to comply with the dialysis schedule and follow-up requirements.
* Patient or his/her legal guardian provides written informed consent.

Exclusion Criteria:

* All contraindications for the EndoForce Connector System according to the IFU.
* Patient is pregnant.
* Patient is enrolled in another dialysis or vascular investigational study, without prior approval from the Sponsor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with end stage renal disease requiring hemodialysis
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2026-01-13 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 2 years
  All device and/or procedure-related events and all major adverse events that reasonably suggest the involvement of the EndoForce and that require or result in any of the following: death, emergent surgery, events requiring hospitalization, events requiring percutaneous interventions, vascular access infection requiring treatment, significant bleeding, pseudoaneurysm and serious adverse events. EndoForce migration, inadequate seal and leakage will also be collected acutely and at each in-person follow-up visit.
AVG Cumulative Patency | 2 years
  The percentage of subjects free from loss of access of the study graft for hemodialysis.
AVG Primary Patency | 2 years
  The percentage of subjects free from the first occurrence of either access thrombosis or an access procedure performed to maintain access patency.
Number of AVG Interventions to Maintain Patency | 2 years
  The number of AVG interventions until access abandonment or through study completion.
Number of Participants with Acute Device Success | Through end of procedure
  AV graft flow at the end of the procedure as determined by palpable graft thrill and/or audible bruit, without significant bleeding or emergent surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Ari Kramer, MD, Principal Investigator — Spartanburg Regional Medical Center
Locations (2):
- United States (2):
  - MUSC Health Orangeburg, Orangeburg, South Carolina
  - Spartanburg Regional Medical Center, Spartanburg, South Carolina

IPD SHARING:
Plan to Share IPD: Yes
IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, CSR